CLINICAL TRIAL: NCT01352520
Title: Phase II Trial of Brentuximab Vedotin (SGN-35) at Dose of 1.8 mg/kg IV Every 3 Weeks in Patients With CD30-positive Lymphoproliferative Disorders (Cutaneous Anaplastic Large T-cell Lymphoma (ALCL), Mycosis Fungoides, and Extensive Lymphomatoid Papulosis (LyP)
Brief Title: SGN-35 in CD30-positive Lymphoproliferative Disorders (ALCL), Mycosis Fungoides (MF), and Extensive Lymphomatoid Papulosis (LyP)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0914; NCI-2011-01045 (Registry Identifier: NCI CTRP-Clinical Trials Registry)
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: CD-30 Positive Anaplastic Large T-cell Cutaneous Lymphoma; Lymphoma, Primary Cutaneous Anaplastic Large Cell; Lymphomatoid Papulosis; Mycosis Fungoides; Skin Lymphoma; Cutaneous Lymphomas; Lymphoma; Hematologic Disorder
Keywords: systemic therapy; cutaneous anaplastic large T cell lymphoma; ALCL; lymphomatoid papulosis; LyP; mycosis fungoides; MF; SGN-35 (brentuximab vedotin); skin lymphomas; CD30-positive lymphoproliferative disorders; tumor lymphocytes; cutaneous lymphomas; CD30+ expression; Hematologic Disorder; Lymphoma
MeSH Terms: conditions — Lymphoma, Primary Cutaneous Anaplastic Large Cell; Lymphomatoid Papulosis; Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous; Lymphoma; Hematologic Diseases | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SGN-35 (Experimental): 1.8 mg/kg intravenously Day 1 of 21-day cycle.
  Interventions: Drug: SGN-35

INTERVENTIONS:
Drug: SGN-35 — 1.8 mg/kg administered by outpatient IV infusion given over approximately 30 minutes on Day 1 of each 21-day cycle.
  Other Names: Brentuximab vedotin

SUMMARY:
The goal of this clinical research study is to learn if SGN-35 (brentuximab vedotin) can help to control ALCL, LyP or MF in patients with at least 1 of the 3 skin lymphomas. The safety of the study drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Brentuximab vedotin is an antibody that is designed to find a certain protein (called CD30) on cancer cells and bind to it. It is designed to then enter the cell and release a molecule that may kill the cancer cells.

Study Drug Administration:

If you are found eligible to take part in this study, you will begin receiving brentuximab vedotin by vein over 30 minutes on Day 1 of each 21-day study cycle. If you have side effects after your first dose and your doctor thinks it is in your best interest, future doses may be lowered or delayed for up to 3 weeks.

Premedications:

If you have any reactions at the infusion site after you receive the study drug during Cycle 1, you may be given acetaminophen (Tylenol) or diphenhydramine (Benadryl) 30-60 minutes before all following infusions.

Study Visits:

At each clinic visit, including follow-up visits (described below), you will have full skin exams. You will be checked to see how much of your skin's surface has lesions. Up to 6 skin lesions will be selected to be photographed and measured at each visit. Your private areas will be covered (as much as possible), and a picture of your face will not be taken unless there are lesions on your face. You will not be able to be identified in the photographs. The following tests and procedures will also be performed:

On Day 1 of all study cycles (before you receive the study drug):

* You will have a physical exam.
* Your performance status will be recorded.
* You will be asked about any drugs that you may be taking and if you are having any side effects.
* You will complete 5 questionnaires about your quality of life and itching symptoms.
* Blood (about 4-6 teaspoons) will be drawn for routine tests and to check the status of the disease.
* If you have not had a lesion biopsy within the last 6 weeks you will have a lesion biopsy to check the status of the disease and for PGx testing.

Length of Study Treatment:

You may receive the study drug for up to 8 cycles. You will be taken off study if the disease gets worse or intolerable side effects occur.

If the disease has a complete response, you may receive the study drug for 2 more cycles if the study doctor thinks it is in your best interest.

If the disease has complete response, then comes back, you may receive the study drug for 8 more cycles if the doctor thinks it is in your best interest.

If you are doing better at the end of 8 cycles but the disease is not in complete remission, the study doctor may allow you to receive the study drug every 3 weeks at the full dose or every 2 weeks at a lower dose for 8 additional cycles. If you continue to have improvement after these 16 cycles, the study doctor may allow you to continue receiving the study drug. The study doctor will discuss this with you.

Follow-up Visits:

About 3-4 weeks after you have stopped taking the study drug, the following tests and procedures will be performed:

* Your medical history will be recorded.
* Your performance status will be recorded.
* You will have a physical exam.
* You will be asked if you are having any side effects.
* You will complete 5 questionnaires about your quality of life and itching symptoms.
* Blood (about 4-6 teaspoons) will be drawn for routine tests and to check the status of the disease.
* You will have a CT or PET scan to check the status of the disease.
* You will have a lesion biopsy to check the status of the disease and for PGx testing.

Long-term Follow-up:

You or your primary doctor may be contacted for long-term follow-up on the status of the disease, any study-related nerve damage (including loss of motor or sensory function) you have, and your overall health status.

Follow-up will be every 12-16 weeks for the first 2 years after the last dose. Then, the follow-up will be every 6 months (+/- 1 month) up to a maximum period of 5 years.

This is an investigational study. Brentuximab vedotin is FDA approved and commercially available for use in patients with ALCL. It is currently being used for LyP and MF for research purposes only. You will receive $15 coupons for valet parking for each clinic visit you make during this study.

Up to 84 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a biopsy confirmed diagnosis based on a combination of histological and clinical criteria of CD30+ lymphomatoid papulosis, CD30+ primary cutaneous anaplastic large T-cell lymphoma (pc-ALCL), or CD30+ mycosis fungoides for the phase II trial. There is no specific limit or validated amount other than positive cells on 1HC cells in tumor cells.
2. Patients with pc-ALCL that has spread systemically (e.g. to lymph nodes, bone marrow or visceral organs) may be included so long as pc-ALCL was the primary diagnosis for at least 6 months before systemic involvement was confirmed. MF patients must be stage IB or greater.
3. Systemic involvement (i.e., nodal, bone marrow or visceral organ involvement) will be evaluated by CT and/or PET and bone marrow biopsy(if indicated on patients with blood involvement) in patients with pc-ALCL or MF at baseline.
4. Patients' biopsies must be histologically confirmed CD30 positive within 36 months of enrollment.
5. pc-ALCL and MF patients must have progressed or relapsed after treatment with local radiation therapy, phototherapy, topical chemotherapy, or have failed systemic therapy of at least one single agent (e.g., methotrexate or bexarotene or other non-CD30 antibody) or one multi-agent chemotherapy (e.g. CHOP: cyclophosphamide, doxorubicin, vincristine, and prednisone). pc-ALCL classified patients are required to have one or more cutaneous tumors that by history have been present for at least 3 months.
6. All patients must be considered an eligible candidate for systemic therapy as determined by the investigator. To be eligible, LYP patients must be in need of systemic therapy ie have scarring or active lesions (>/=10 per month), or any number of active lesions on face, hands or feet.
7. Patients must have the following minimum wash-out from previous treatments: a. >/= 4 weeks for local radiation therapy, systemic cytotoxic anticancer therapy, treatment with other anticancer investigational agents. b. > 2 weeks for oral methotrexate, retinoids or biological response modifiers therapy for any indication, or topical prescription or topical therapy. c. >/= 12 weeks for any immunotherapy (e.g., monoclonal antibody). Patients with rapidly progressive disease may be treated earlier than the required washout period; patients should have recovered from prior treatment-related toxicities
8. Patients must have an ECOG performance status of </= 2.
9. Patients must be at least 18 years of age.
10. Patients must be available for periodic blood sampling, study-related assessments, and management of toxicity at the treating institution.
11. Females of childbearing potential [a female not post menopausal for at least 12 months or not surgically sterilized] must have a negative beta-HCG pregnancy </=7 days prior to Day 1 of Cycle 1. If the pregnancy test is outside institutional normal range at pretreatment, the subject must have a second pregnancy test. If the second pregnancy test is outside institutional normal range then a gynecology consult is needed to confirm the subject is not pregnant. All patients must agree to use an effective contraceptive method during the course of the study.
12. Patients must give written informed consent. A copy of the signed informed consent form will be retained in the patient's chart.
13. The following required baseline laboratory data: absolute neutrophil count (ANC) >/= 1000/microliter, platelets >/= 50,000/µL (unless documented bone marrow involvement with lymphoma), bilirubin </= 1.5X upper limit of normal (ULN) or </= 3X ULN for patients with Gilbert's disease, serum creatinine </= 1.5X ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 2.5X ULN.

Exclusion Criteria:

1. Concomitant corticosteroid use for systemic or topical treatment of skin disease is not allowed except a dose of steroid of no more than 20 mg of prednisone or its equivalence is allowed of asthma, COPD or IBD .Stable use of topical corticosteroids of mid-potency will be allowed for patients with erythroderma-Sezary syndrome (T4) and tumor stage (T3) with intense pruritus.
2. Patients with known grade 3 or higher (per CTCAE v.4.0 criteria) active systemic or cutaneous viral, bacterial or fungal infection.
3. Patients who are known to be HIV, Hepatitis B, or Hepatitis C positive.
4. Patients with known hypersensitivity to recombinant proteins or any excipient contained in the drug formulation that includes trehalose, sodium citrate, and polysorbate 80.
5. Patient with a history of other malignancies during the past three years. (The following are exempt from the 3-year limit: non-melanoma skin cancer, melanoma in situ, curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on PAP smear.)
6. Patients with congestive heart failure, Class III or IV, by the NYHA criteria.
7. Patients who are pregnant or breastfeeding.
8. Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment.
9. Patients with dementia or altered mental status that would preclude understanding and rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 12 months
  Response rate is percentage of participants with skin lesions that express CD30+ receiving SGN-35 in primary cutaneous ALCL, MF, and extensive lymphomatoid papulosis whose best response during the observation period is a Partial Response (PR), regression of measurable disease, or Complete Response (CR), complete disappearance of all clinical evidence of disease, (i.e. at least moderate improvement). Objective tumor response (PR, CR, PR+CR) based on Response Evaluation Criteria In Solid Tumors (RECIST) criteria.

SECONDARY OUTCOMES:
Time to Progression | Assessments through 8 treatment cycles (21 day cycle, approximately 6 months) with possible expansion to 16 cycles, up to 2 years.
  Time to progression calculated as the time (days) from date of first dose of study drug to date of first observed progression or death date if the death was due to disease progression whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Auris O Huen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lewis DJ, Talpur R, Huen AO, Tetzlaff MT, Duvic M. Brentuximab Vedotin for Patients With Refractory Lymphomatoid Papulosis: An Analysis of Phase 2 Results. JAMA Dermatol. 2017 Dec 1;153(12):1302-1306. doi: 10.1001/jamadermatol.2017.3593. PMID 28980004
- See also: M D Anderson Cancer Center — http://www.mdanderson.org